CLINICAL TRIAL: NCT04326153
Title: A Single-center Phase 2 Study of Neoadjuvant Immunotherapy Plus Chemotherapy for Potentially Resectable Stage IIIA/IIIB Non-Small Cell Lung Cancer
Brief Title: Neoadjuvant Immunotherapy Plus Chemotherapy for Potentially Resectable Stage IIIA/IIIB Non-Small Cell Lung Cancer
Acronym: Neo-Pre-IC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2019158
Record Dates: First submitted 2020-03-17; First posted 2020-03-30 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-12

CONDITIONS: IIIA Stage Non-small Cell Lung Cancer
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental arm (Experimental): Sintilimab+Albumin paclitaxel:+Carboplatin:
  Interventions: Drug: Sintilimab Injection

INTERVENTIONS:
Drug: Sintilimab Injection — Preoperative:
  Sintilimab: 200mg QD, one cycle every 21 days, the first day of each cycle, a total of two cycles.
  Albumin paclitaxel: 135mg / m2 QD, 1 cycle every 21 days, 1 day and 8 days of each cycle, 2 cycles in total.
  Carboplatin: AUC 5mg QD, one cycle every 21 days, two cycles in total
  Postoperative:
  Patients began to receive postoperative adjuvant treatment within 21-60 days after the operation. Specific medication plan:
  Sintilimab: 200mg QD, one cycle every 21 days, the first day of each cycle, a total of 8 cycles.
  Albumin paclitaxel: 135mg / m2 QD, 1 cycle every 21 days, 1 day and 8 days of each cycle, 2 cycles in total.
  Carboplatin: AUC 5mg QD, one cycle every 21 days, two cycles in total.

SUMMARY:
Cancer has always been one of the leading causes of death in the world, and China is facing more and more severe challenges from cancer. Among all the causes of cancer death, lung cancer (25.2%) ranks first, among which non-small cell lung cancer (NSCLC) accounts for about 80% to 85%, of which about 1 / 3 of the patients have been in the local advanced stage (IIIA stage / IIIB stage) at the time of initial diagnosis. For the patients with stage IIIA NSCLC who can be operated on, surgery is still the most effective way to treat them. Even so, NSCLC in stage I-III undergoing radical surgery is the most effective way 30-60% of the patients eventually had relapse or distant metastasis. Therefore, people began to explore a new treatment mode, preoperative neoadjuvant chemotherapy, to improve the survival rate of NSCLC 2.

At present, the NCCN guidelines for the new adjuvant treatment of NSCLC mainly recommend platinum based dual drug chemotherapy.

Immunotherapy combined with chemotherapy will be a potential new adjuvant therapy in the future, which can improve the resection rate of patients, reduce the recurrence rate after surgery, and have tolerable adverse reactions.

DETAILED DESCRIPTION:
Sample size calculation： The primary endpoint is the 2-year DFS rate，however, due to the extended observation time required for this endpoint, it is not suitable for promptly validating treatment response. MPR rate is employed to calculate the necessary sample size.

Simon's optimal two-stage design is utilized. The addition of sintilimab to chemotherapy is assumed to elevate the MPR rate from 8.9% to 35%. The sample size should be 29(17+12). In the first stage, the study will be concluded if ≤2 patients achieve MPR, indicating a negative outcome. Conversely, if more than 4 patients achieve MPR, the study will proceed by enrolling an additional 12 patients. Considering the sample size calculation results and sufficient funding, the final enrollment is 30. The type 1 error rate is 0.05. The outlined protocol yield an 95% statistical power to detect an MPR rate of 35% under alternative hypotheses.

MRD detectition： Using previously retained biomarkers from patients for MRD detection, exploring the relationship between MRD and patient DFS and OS.

ELIGIBILITY:
Inclusion Criteria:

1. Asian male or female patients: 18-75 years old;
2. ECoG physical condition score: 0-2;
3. Histologic examination confirmed that the potential resectable stage IIIA/IIIB non-small cell lung cancer (T4 or N2 according to the TNM staging standard of AJCC 8th Edition);
4. Estimated survival time ≥ 12 weeks;
5. No systemic anti-tumor therapy has been received before. The function of main organs is normal, that is to say, the relevant examination indexes within 14 days before randomization meet the following requirements:

1) Blood routine examination:

a) Hemoglobin ≥ 90 g / L (no blood transfusion within 14 days); b) Neutrophil count ≥ 1.5 × 109 / L; c) Platelet count ≥ 100 × 109 / L;

2) Biochemical examination:

a) Total bilirubin ≤ 1.5 × ULN (upper limit of normal value); b) ALT or AST ≤ 2.5 × ULN; ALT or AST ≤ 5 × ULN in case of liver metastasis; c) Serum creatinine < 1.5 times of the upper limit of normal value; endogenous creatinine clearance ≥ 50 ml / min (Cockcroft Gault formula);

3) Routine coagulation examination:

1. INR or PT ≤ 1.5 x ULN.
2. APTT ≤ 1.5 x ULN.

   4) Left ventricular ejection fraction (LVEF) ≥ 50%.

   7. Pregnant women of childbearing age must carry out pregnancy test (serum or urine) within 7 days before entering the group, and the result is negative, and they are willing to use appropriate methods of contraception during the test and within 8 weeks after the last administration of the test drug. For men, it is necessary to agree to use appropriate methods of contraception or sterilization after operation during the trial period and within 8 weeks after the last administration of the test drug;

   8. Good compliance, family members agree to cooperate to receive survival follow-up;

   9. Sign informed consent.

   Exclusion Criteria:
   1. There are mixed small cell carcinoma and sarcoma in histology;
   2. Other malignant tumors were diagnosed within 5 years before administration, excluding radical skin basal cell carcinoma, skin squamous cell carcinoma and / or radical resection of carcinoma in situ. If more than 5 years before the administration of the drug is diagnosed as other malignant tumors or lung cancer, it is necessary to carry out pathological or cytological diagnosis of the recurrent lesions;
   3. Currently participating in the intervention clinical research and treatment, or receiving other drugs or research instruments within 4 weeks before the first administration;
   4. Previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs for another stimulation or synergistic inhibition of T cell receptor (such as CTLA-4, OX-40, CD137);
   5. Received immunomodulatory drugs (thymosin, interferon, interleukin, etc.) within 2 weeks before the first administration, or received major surgical treatment within 3 weeks before the first administration;
   6. With a history of haemorrhagic disease, any bleeding event with a severe grade of 3 or more in ctcae5.0 occurred within 4 weeks before screening;
   7. Received solid organ or blood system transplantation;
   8. There are clinically uncontrolled active infections, including but not limited to acute pneumonia;
   9. There were idiopathic pulmonary fibrosis, organic pneumonia (such as bronchiolitis obliterans), and drug-related pneumonia;
   10. Uncontrollable or symptomatic hypercalcemia;
   11. III-IV and congestive heart failure (New York Heart Association classification), poorly controlled and clinically significant arrhythmias;
   12. It is known to have allergic reactions to PD-1 monoclonal antibody, albumin paclitaxel, carboplatin active ingredients and / or any excipients;
   13. Active autoimmune diseases requiring systemic treatment (e.g., use of disease improving drugs, corticosteroids or immunosuppressants) occurred within 2 years before the first administration. Alternative therapies (such as thyroxine, insulin or corticosteroids in physiological doses for adrenal or pituitary insufficiency) are not considered systemic.
   14. Patients who need long-term systemic corticosteroid use. Patients with COPD, asthma requiring intermittent use of bronchodilators, inhaled corticosteroids, or local injection of corticosteroids were included.
   15. Long term unhealed wound or incomplete union fracture;
   16. Active infection requiring treatment or systemic anti infective drugs used within 1 week before the first administration;
   17. In the first 6 months of screening, there were arterial thrombosis events, such as cerebrovascular accident (including transient ischemic attack), myocardial infarction, unstable angina, etc;
   18. For female subjects: they should be surgical sterilization, postmenopausal patients, or agree to use a medically recognized contraceptive measure during the study treatment period and within 6 months after the end of the study treatment period; the serum or urine pregnancy test must be negative within 7 days before the study is enrolled in the group, and must be non lactation period. Male subjects: patients who should be sterilized surgically or who agree to use a medically approved contraceptive method during the study and within 6 months after the end of the study.
   19. Known human immunodeficiency virus (HIV) infection history (i.e. HIV 1 / 2 antibody positive);
   20. Untreated active hepatitis B;

       Note: hepatitis B subjects who meet the following criteria also meet the inclusion criteria:

       Before the first administration, HBV viral load must be less than 1000 copies / ml (200iu / ml). Subjects should receive anti HBV treatment during the whole period of chemotherapy drug treatment to avoid virus reactivation. For subjects with anti HBC +, HBsAg (-), anti HBS (-), and HBV viral load (-), prophylactic anti HBV treatment is not required, but virus reactivation needs to be closely detected.
   21. Active HCV infected subjects (HCV antibody positive and HCV-RNA level higher than the detection limit)
   22. Those who have a history of abuse of psychotropic substances and are unable to give up or have mental disorders;
   23. Inoculate the live vaccine within 30 days before the first administration; Note: it is allowed to receive the injection inactivated virus vaccine for seasonal influenza; however, it is not allowed to accept the live attenuated influenza vaccine for intranasal medication.

   There are medical history, disease, treatment or laboratory abnormal results that may interfere with the test results, prevent the subjects from participating in the whole process of the study, or the researchers think that participating in the study is not in the best interests of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
2 years DFS rate | 2 years
  To evaluate the 2-year DFS rate of neoadjuvant treatment of Asian patients with resectable stage IIIA NSCLC with Sintilimab combined with albumin paclitaxel and carboplatin

SECONDARY OUTCOMES:
MPR rate | 36 month
  Major pathological remission rate
PCR rate | 36 month
  Pathological complete response rate
Downgrade rate | 36 month
  Downgrade rate,including T downgrade and N downgrade
DFS | 36 month
  Disease-free survival
OS | 36 month
  Overall survival
ORR | 36 month
  Objective response rate
TRAE | 36 month
  Treatment-related adverse reactions

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital Of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No